CLINICAL TRIAL: NCT06189859
Title: Electrosurgical Modes for Endoscopic Submucosal Dissection in Peroral Endoscopic Esophageal Myotomy: a Randomized Controlled Trial
Brief Title: Electrosurgical Modes for Endoscopic Submucosal Dissection in Peroral Endoscopic Esophageal Myotomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Shehab, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESRCT
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Achalasia; Achalasia Cardia
Keywords: achalasia; POEM; ELECTROSURGERY; SPRAY COAGULATION; PERORALENDOSCOPIC ESOPHAGEAL MYOTOMY
MeSH Terms: conditions — Esophageal Achalasia; Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation of patients will be in sealed envelopes to be opened on day of the procedure. The investigator and care provider (same) will thus be unmasked. Participant and outcomes assessor will remain masked until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spray coag mode (Active Comparator): After initial mucosal incision, Endoscopic submucosal dissection will be performed using Spray coag mode using ERBE VIO 3 generator (effect 3-3.5)
  Interventions: Procedure: endoscopic submucosal dissection using SPRAY COAG mode
- Precisect mode (Active Comparator): After initial mucosal incision, Endoscopic submucosal dissection will be performed using Precisect mode using ERBE VIO 3 generator (effect 4.5-5)
  Interventions: Procedure: endoscopic submucosal dissection using Precisect mode

INTERVENTIONS:
Procedure: endoscopic submucosal dissection using SPRAY COAG mode — After initial mucosal incision, submucosal dissection will be performed down to 2cm below the cardia using Spray coag mode using ERBE VIO3 generator and a Hybrid knife (T-type) aided by ERBEJET for submucosal injection
  Other Names: POEM
  Arms: Spray coag mode
Procedure: endoscopic submucosal dissection using Precisect mode — After initial mucosal incision, submucosal dissection will be performed down to 2cm below the cardia using Precisect mode using ERBE VIO3 generator and a Hybrid knife (T-type) aided by ERBEJET for submucosal injection
  Arms: Precisect mode

SUMMARY:
Peroral endoscopic esophagel myotomy (POEM) is a third space endoscopy technique that depends on creating a submucosal tunnel to expose the esophageal muscle and eventually perform an esophageal myotomy. Submucosal dissection can be performed using numerous electrosurgical modes. Spray coagulation has been anecdotally favored by many endoscopists due to its high coagulation power and assumed safety. Recently, Precisect mode has been developed, it has theoretical advantages of very minimal tissue penetration and minimal to no charring effect. In this trial, the investigators compare the efficacy and safety of both electrosurgical modes in POEM procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing POEM procedure for any esophageal motility disorder
* Esophageal motility disorder confirmed by high-resolution manometry and gastroscopy

Exclusion Criteria:

* Esophageal varices
* Esophageal neoplasms
* Non-correctable coagulopathy
* Failure to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Speed of endoscopic submucosal dissection | during the procedure
  Speed of dissection (cm/minute)

SECONDARY OUTCOMES:
Intraprocedural Bleeding | during the procedure
  Bleeding necessitating change in electrosurgical mode
Significant Intraprocedural bleeding | during the procedure
  Bleeding necessitating change of instrument to coagulating forceps
Other Adverse events | during the procedure
  Including mucosal injury, postoperative pain, postoperative bleeding and other complications
Total procedure duration | during the procedure
  Total procedure duration
Endoscopic submucosal tunneling duration | during the procedure
  Endoscopic submucosal tunneling duration

CONTACTS AND LOCATIONS:
Overall Officials: hany shehab, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No